CLINICAL TRIAL: NCT05637775
Title: DiSCIoser: Unlocking Recovery Potential of Arm Sensorimotor Functions After Spinal Cord Injury by Promoting Activity-dependent Brain Plasticity and Modeling the Causal Relationship Between Brain Plasticity and Recovery of Function
Brief Title: DiSCIoser: Improving Arm Sensorimotor Functions After Spinal Cord Injury Via Brain-Computer Interface Training
Acronym: DiSCIoser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Donatella Mattia, Professor, Laboratory Director, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2019-12369396
Record Dates: First submitted 2022-11-21; First posted 2022-12-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Motor Disorders
Keywords: spinal cord injury; brain computer interface; motor imagery; motor rehabilitation; neurorehabilitation; brain plasticity
MeSH Terms: conditions — Spinal Cord Injuries; Motor Disorders

STUDY DESIGN:
Intervention Model Description: Eligible subacute cervical SCI patients admitted to Fondazione Santa Lucia Hospital for standard rehabilitation care will be randomized in equal proportions (1:1 ratio) between BCI-assisted MI training- EXP) and Control (MI without BCI - CTRL).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors performing clinical evaluation and data analysts will be blinded to patient allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXP - BCI (Experimental): (EEG-)BCI- assisted MI training delivered as add-on regimen (Standard physiotherapy-3 h/day, 5 day/week).
  Interventions: Other: EEG-based BCI system for (hands) Motor Imagery training
- CTRL - MI (Active Comparator): MI training delivered as add-on regimen (Standard physiotherapy-3 h/day, 5 day/week).
  Interventions: Other: Control - MI intervention

INTERVENTIONS:
Other: EEG-based BCI system for (hands) Motor Imagery training — For the purposes of this study we adapted an available BCI-supported motor imagery (MI) training station, equipped with a computer, a commercial wireless Electroencephalography (EEG)/ Electromyography (EMG) system, a screen for therapist feedback and a screen for the real-time ecological feedback to patient - a custom software program that provides a for (personalized) visual representation of the patient's own hands. This software allows the therapists to create an artificial reproduction of patient's hands/forearms by adjusting a digitally created image in shape, size, skin colour and orientation to match as much as possible the real patient hands/forearms. Training consists of the MI tasks of both hands, grasping or finger extension in separate runs. The trial length will include a constant baseline period of 4 sec and a task period of maximally 10 sec for BCI intervention group. Each training session will consist of 4 runs (20 trials each).
  Other Names: BCI - EXP
  Arms: EXP - BCI
Other: Control - MI intervention — Training consists of MI tasks of both hands, grasping or finger extension in separate runs. MI training will be delivered with a dose/setting regimen equivalent to EXP intervention. The trial length will include a constant baseline period of 4 sec and a task period of maximally 4 sec. Each training session will consist of 4 runs (20 trials each).
  Other Names: MI - CTRL
  Arms: CTRL - MI

SUMMARY:
The goal of this clinical trial is to validate the efficacy of a Brain-Computer Interface (BCI)-based intervention for hand motor recovery in subacute cervical spinal cord injured (SCI) patients during rehabilitation. The study will provide evidence for the clinical/neurophysiological efficacy of the BCI intervention as a means to promote cortical sensorimotor plasticity (remote plasticity) and thus maximize recovery of arm functions in subacute cervical SCI. Participants will undergo an extensive clinical, neurophysiological, neuropsychological and neuroimaging assessment before and after a BCI training based on motor Imagery (MI) of hands. The intervention will be delivered with a system that was originally validated for stroke patients and adapted to the aims of this study. Researchers will compare the BCI intervention with an active MI training without BCI support (active comparator).

DETAILED DESCRIPTION:
Despite its relatively low incidence SCI represents a devastating chronic condition for which there is still no cure or consistent approach for intervention. Cervical SCI tremendously affects the quality of life since the use of the upper extremities is critical for completing basic activities of daily living. Extensive research conducted on SCI animal models and humans has revealed that cortical and subcortical reorganization (ie., remote plasticity) takes place after SCI and it is associated with recovery of sensorimotor function (in humans the relevance of these aspect has been mainly emphasised in incomplete SCI). Current rehabilitation after traumatic SCI mainly consists of intensive training of lost/impaired function that is assumed to augment activity-dependent plasticity of spared circuits and thus, leading to functional improvements. Recently, neuromodulatory interventions targeting the sensorimotor systems at various levels has been applied in humans with SCI in combination with training to enhance functional recovery. Neurological rehabilitation of SCI can also benefit of cognitive training based on MI, that enables active stimulation of brain motor areas promoting brain plasticity associated with positive effects on motor performance. In the effort of encouraging the top-down contribution of supraspinal sensorimotor signaling in SCI rehabilitation, the BCI technology may provide for fundamental tools not only for restoring but even recovering sensorimotor function. The long history of BCI research in SCIs has been substantially devoted to develop systems to control external devices to restore function. However, recent findings indicate that non invasive BCI training in combination with intensive rehabilitation can be beneficial to chronic SCI patients for gait, as well as arm function recovery. The current study relies on the hypothesis that monitoring and modulating brain plasticity occurring as a consequence of a SCI is a key factor in shaping clinically valuable top-down rehabilitation strategies that target the recovery of sensorimotor function in patients with SCI. To ground such vision, the researchers will use a goal-oriented action imagery training which is controlled and objectified by a BCI as a means to engage sensorimotor system and thus to facilitate neuroplasticity and optimize functional recovery in SCI during the subacute phase in which brain and spinal plasticity is at its climax.

In this study researchers will test the superiority of a BCI-assisted MI training (up to 12 weeks duration) with respect to MI practiced without BCI feedback (similar training setting and duration) to promote recovery of sensorimotor functions in traumatic cervical SCI subjects. The main hypothesis is that establishing a real-time contingency between the content of MI and an ecological feedback specifically designed to train MI in SCI patients will boost the effect of MI training in engaging the sensorimotor system. Primary and secondary outcome measures (reported in the dedicated section) include the most commonly used clinical and functional scales to assess SCI patients recovery. Neurophysiological and Neuroimaging outcomes are reported as other outcome measures in the dedicated session. Neuropsychological evaluation will include Test of Attentional Performance (TAP), Stroop Test, Trail Making Test (TMT), assessment of depression and anxiety; body ownership and representation. Furthermore, motivation, satisfaction, workload and usability will be evaluated along training.

ELIGIBILITY:
Inclusion Criteria:

* subacute cervical SCI (30-90 days from event)
* classification according to ISNCSCI AIS A-D, lesion level C1-T1
* Upper Extremity Motor Score (UEMS) < 40

Exclusion Criteria:

* other conditions (present or previous) potentially affecting sensorimotor upper limb function
* inability to give informed consent and understand the requirements for the training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline on Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) somatosensory scores of bilateral arms at end of intervention | Pre-Randomization, Post Training (within 48 hours)
  The GRASSP scale (somatosensory sub-section) ranges from 0 (maximum impairment) to 12 (normal) for each side arm.

SECONDARY OUTCOMES:
Mean change from baseline on Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) motor scores of bilateral arms at end of intervention | Pre-Randomization, Post Training (within 48 hours)
  The GRASSP scale (motor sub-section) ranges from 0 (maximum impairment) to 50 (normal) for each side arm.
Mean change from baseline in the Spinal Cord Injury Independence Measure (SCIM) - self care section | Pre-Randomization, Post Training (within 48 hours)
  The SCIM is the most commonly used independence scale for SCI patients. The Self Care section includes questions on feeding, grooming, bathing and dressing ranging from 0 (dependence) to 20 (independence).
Mean change in Pain as assessed by the International SCI Pain Basic Dataset (ISCIPBDS) | Pre-Randomization, Post Training (within 48 hours)
  The ISCIPBDS assesses pain in SCI patients. The questions concern pain severity, physical and emotional function and include a pain-intensity rating, a pain classification and questions related to the temporal pattern of pain for each specific pain problem. The impact of pain on physical, social and emotional function, and sleep is evaluated for each pain. Each question ranges from 0 to 10.
Mean change in Upper Extremity Motor Score (UEMS) from the ISNCSCI AIS evaluation | Pre-Randomization, Post Training (within 48 hours)
  The UEMS of the AIS assessment evaluates residual strength in upper limb segments and ranges from 0 to 50 (for both arms)

OTHER OUTCOMES:
Changes from baseline on high density Electroencephalography (hdEEG) patterns of cortical oscillatory activity and connectivity at end of intervention. | Pre-Randomization, Post Training (within 1 week)
  EEG recordings (motor relevant oscillatory activity and functional connectivity at rest and task related) to evaluate the neurophysiological substrates of the experimental intervention efficacy, in both BCI-based and Control intervention groups at end of treatment.
Changes in Motor Evoked Potentials (MEPs) | Pre-Randomization, Post Training (within 1 week)
  MEPs elicited via Transcranial Magnetic Stimulation (TMS) to evaluate the integrity of the Cortico Spinal Tract (CST) in both experimental and Control groups as factor influencing experimental intervention response
Changes in Somatosensory Evoked Potentials (SSEPs) | Pre-Randomization, Post Training (within 1 week)
  SSEPs from upper and lower limb nerves and recorded at peripheral and central stations via surface electrodes.
Structural Magnetic Resonance Imaging (MRI) of the whole brain and spinal cord | Pre-Randomization, Post Training (within 1 week)
  structural MRI to evaluate lesion size/site at the spinal cord level and cortico-spinal tract integrity in both experimental and Control groups as factor influencing experimental intervention response

CONTACTS AND LOCATIONS:
Overall Officials: Donatella Mattia, MD, PhD, Principal Investigator — Fondazione Santa Lucia, IRCCS; Giorgio Scivoletto, MD, PhD, Principal Investigator — Fondazione Santa Lucia, IRCCS; Febo Cincotti, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Neurorehabilitation Units- Fondazione Santa Lucia, IRCCS, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Clinical, Neurophysiological, Neuropsychological and Neuroimaging Data will eventually be shared upon reasonable request (anonymized)

REFERENCES:
- [Background] Pichiorri F, Morone G, Petti M, Toppi J, Pisotta I, Molinari M, Paolucci S, Inghilleri M, Astolfi L, Cincotti F, Mattia D. Brain-computer interface boosts motor imagery practice during stroke recovery. Ann Neurol. 2015 May;77(5):851-65. doi: 10.1002/ana.24390. Epub 2015 Mar 27. PMID 25712802
- [Background] Donati AR, Shokur S, Morya E, Campos DS, Moioli RC, Gitti CM, Augusto PB, Tripodi S, Pires CG, Pereira GA, Brasil FL, Gallo S, Lin AA, Takigami AK, Aratanha MA, Joshi S, Bleuler H, Cheng G, Rudolph A, Nicolelis MA. Long-Term Training with a Brain-Machine Interface-Based Gait Protocol Induces Partial Neurological Recovery in Paraplegic Patients. Sci Rep. 2016 Aug 11;6:30383. doi: 10.1038/srep30383. PMID 27513629
- [Background] Brown AR, Martinez M. From cortex to cord: motor circuit plasticity after spinal cord injury. Neural Regen Res. 2019 Dec;14(12):2054-2062. doi: 10.4103/1673-5374.262572. PMID 31397332
- [Background] Mattia D, Pichiorri F, Colamarino E, Masciullo M, Morone G, Toppi J, Pisotta I, Tamburella F, Lorusso M, Paolucci S, Puopolo M, Cincotti F, Molinari M. The Promotoer, a brain-computer interface-assisted intervention to promote upper limb functional motor recovery after stroke: a study protocol for a randomized controlled trial to test early and long-term efficacy and to identify determinants of response. BMC Neurol. 2020 Jun 27;20(1):254. doi: 10.1186/s12883-020-01826-w. PMID 32593293
- [Derived] Colamarino E, Lorusso M, Pichiorri F, Toppi J, Tamburella F, Serratore G, Riccio A, Tomaiuolo F, Bigioni A, Giove F, Scivoletto G, Cincotti F, Mattia D. DiSCIoser: unlocking recovery potential of arm sensorimotor functions after spinal cord injury by promoting activity-dependent brain plasticity by means of brain-computer interface technology: a randomized controlled trial to test efficacy. BMC Neurol. 2023 Nov 21;23(1):414. doi: 10.1186/s12883-023-03442-w. PMID 37990160